CLINICAL TRIAL: NCT00989768
Title: Field Effects of Two Commercial Preparations of Botulinum Toxin Type a Administered to the Frontalis Muscles
Brief Title: Field of Effects of Two Commercial Preparations of Botulinum Toxin Type A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Doris Hexsel, CBED
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-CBED06b
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2010-04-27 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-10

CONDITIONS: Wrinkles in Frontal Area
Keywords: Botulinum toxin type A; field effects; dose-equivalence; anhydrotic action halos
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum toxin type - A (Experimental): Dysport® compared to Botox®
  Interventions: Drug: Botulinum Toxin Type A (Dysport®); Drug: Botulinum Toxin Type A/Botox®; Drug: Botulinum Toxin Type A/Dysport®

INTERVENTIONS:
Drug: Botulinum Toxin Type A (Dysport®) — Botulinum toxin A (Dysport®)will be administered according to an equivalence ratio of 2,5:1. Both reconstituted in the same volume per point, injected in the forehead determined site.
  -Dysport®: 5 units will be injected in the left or right forehead side.
Drug: Botulinum Toxin Type A/Botox® — 2 units will be injected in the left or right forehead side.(opposite side of dysport injection)
Drug: Botulinum Toxin Type A/Dysport® — Botulinum toxin A (Dysport®)will be administered according to an equivalence ratio of 2:1. Both reconstituted in the same volume per point, injected in the forehead determined site.
  -Dysport®: 4 units will be injected in the left or right forehead side, 2:1 ratio Dysport/Botox.

SUMMARY:
The objective of this study is to compare the field of effects of the botulinum toxins (Dysport® and Botox®) using two equivalence-ratios and to gather supportive information, such as more detailed data on the effectiveness in reduction of wrinkles and duration of action on the upper part of the face of both products, trough scales and photographs evaluations.

DETAILED DESCRIPTION:
This was a monocentric, prospective, randomized and double-blind study. Twenty nine female patients, presenting with moderate to severe forehead wrinkles, with sweating ability who had never undergone previous BoNT-A injections were enrolled. Subjects have received botulinum toxin type-A injections in two forehead sites, Botox 2U and Dysport 5U, both reconstituted in the same volume of 0.02 mL per point. Baseline, twenty-eight and 112 days later, clinical and photographic assessments, Minor´s test, and electromyographic (EMG) evaluations were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent (Annex 1)
2. Female
3. Subjects agreeing to take part in all procedures of the study, including botulinum toxin applications, Minor's test, measurement of Evoked Potentials, photographs, etc.), after being fully informed on the objectives and nature of the investigations
4. Subjects aged between 18 and 60 years
5. Subjects presenting with moderate to severe wrinkles on the forehead under maximum voluntary contraction of the m. frontalis
6. Subjects with positive Minor's test showing sweating on the forehead in standardized conditions described in Annex 2

   *The Minor's Test will be the last inclusion criterion to be evaluated. Only these patients eligible according to the other inclusion criteria will undergo the Minor's Test to evaluate their sweating on the forehead. The cut off point is a positive Minor's Test (Level +1) - only subjects with Minor's Test (Level +1) will be recruited in the study (Annex 2).
7. Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the products under investigation
8. Subjects of childbearing age should present a negative urine pregnancy test at baseline and should be using an effective contraceptive method;
9. Availability of the patient throughout the duration of the study (112 days)
10. Subject agrees not to undergo other cosmetic or dermatological procedures during the study
11. Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by this protocol

Exclusion Criteria:

1. Pregnant women or women intending to become pregnant in the next 4 months after screening for eligibility
2. Subjects who are lactating
3. Subjects having undergone botulinum toxin treatment within the last 6 months
4. Subjects participating in other clinical trials
5. Any prior surgery affecting the frontalis and/or orbicularis muscles, prior blepharoplasty or brow lift
6. Any prior cosmetic procedures, including fillers, or scars that may interfere with the study results
7. Subjects presenting fronto-parietal alopecia according to the Norwood-Hamilton classification
8. Subjects with neoplastic, muscular or neurological diseases
9. Subjects using aminoglycoside and penicillamine antibiotics, quinine and Ca2+ channel blockers
10. Subjects with inflammation or active infection in the area to be injected
11. Subjects presenting evident facial asymmetry
12. Subjects with a history of adverse effects, such as sensitivity to the components of the formula, ptosis or any other adverse effect, which in the investigator's opinion should prevent the patient from participating in the study
13. Subjects presenting myasthenia gravis, Eaton-Lambert Syndrome and motor neuron diseases
14. Subjects with coagulation disorders or using anticoagulants
15. Subjects with known systemic autoimmune diseases
16. Subjects with a history of medical treatment non-adherence or showing unwillingness to adhere to the study protocol
17. Any condition that, in the opinion of the investigator, can compromise the evaluation of the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator
Locations (1):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 29 subjects was recruited at Brazilian Center For Studies in Dermatology, in Porto Alegre, Brazil. The anticipated drop out rate is 10%. Participants were their own control, because on one side of frontal region they have received 5U of botulinum toxin - Dysport and on other side 4U of botulinum toxin - Botox;
Pre-assignment Details: 13 volunteers were excluded; Screen failure: Iodine allergy = 2; Minor´s Test failure = 6 Mild wrinkles = 3 Inclusion criteria failure = 2
  Minor's test allows the visualization of the area covered by the effects of botulinum toxin on sweat glands also known as action halos.
Groups:
- Dysport® 5U/ Botox® 2U: Botulinum toxin A (Dysport®) 5 U Subjects have received one injection of five units of botulinum toxin , called Dysport® on one side in the frontal region, that the other brand Botox® was administered two units to the other side of the frontal region.
Period: Overall Study
Arm/Group | Dysport® 5U/ Botox® 2U
Started | 29 (All patients received both treatments. They are their own controls)
Completed | 28
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dysport® 5U/ Botox® 2U
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Horizontal Action Halo Diameter at 28 Days
Description: The colorful complex formed by Minor's test allows the visualization of the area covered by the effects of botulinum toxin on sweat glands, also known as action halos. The horizontal diameter at day 28 were expressed in centimeters and quantified by the software Mirror® (Canfield Scientific Inc., USA).
Time Frame: 28 Days
Measure: Mean (Standard Deviation); unit: centimeter
Groups:
- Dysport® 5U: Botulinum toxin A (Dysport®) 5 U Subjects have received one injection of five units of botulinum toxin , called Dysport® on one side in the frontal region.
- Botox® 2U: Two units of Botox® was administered to the other side of the frontal region.
Arm/Group | Dysport® 5U | Botox® 2U
Number analyzed (Participants) | 28 | 28
centimeter | 1.28 (0.26) | 1.12 (0.31)
Statistical Analysis 1: Comparison: Dysport® 5U vs Botox® 2U; In this study the null hypothesis was that BoNT-A1 had the same effect (halus)than the BoNT-A2; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean Difference (Net) = 0.16, Standard Deviation 0.36

2. Primary Outcome: Horizontal Action Halo Diameter at 112 Days
Description: The colorful complex formed by Minor's test allows the visualization of the area covered by the effects of botulinum toxin on sweat glands, also known as action halos. The horizontal diameter at day 112 were expressed in centimeters and quantified by the software Mirror® (Canfield Scientific Inc., USA).
Time Frame: 112 days
Measure: Mean (Standard Deviation); unit: centimeter
Groups:
- Dysport® 5U: Subjects have received one injection of five units of botulinum toxin , called Dysport® on one side in the frontal region.
Arm/Group | Dysport® 5U | Botox® 2U
Number analyzed (Participants) | 28 | 28
centimeter | 1.12 (0.26) | 0.96 (0.29)
Statistical Analysis 1: Comparison: Dysport® 5U vs Botox® 2U; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

3. Secondary Outcome: ECMAP in m. Frontialis
Description: The measurement of the ECMAP(Evoked Compound Muscle Action Potentials) used surface electrodes on the forehead and electrical stimulation of the facial nerve, according to standard neurophysiological procedures. The amplitude of the ECMAP in the m. frontalis on stimulation of the facial nerve was performed by an experienced neurologist. ECMAP was assessed by an electromyography (EMG) device (TECA Sapphire - TECA Corp., Pleasantville, NY).
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Botox ® 2U: Two units of Botox® was administered to the other side of the frontal region.
Arm/Group | Dysport® 5U | Botox ® 2U
Number analyzed (Participants) | 28 | 28
microvolts | 492.53 (290.70) | 468.27 (263.31)
Statistical Analysis 1: Comparison: Dysport® 5U vs Botox ® 2U; Test type: Superiority or Other; p = 0.61, t-test, 2 sided

4. Secondary Outcome: ECMAP in m. Frontialis
Description: as for outcome 3
Time Frame: 112 days
Measure: Mean (Standard Deviation); unit: microVolts
Groups:
- Botox® 2U: Two units of Botox® was administered two units to the other side of frontal region
Arm/Group | Dysport® 5U | Botox® 2U
Number analyzed (Participants) | 28 | 28
microVolts | 482.63 (279.58) | 539.16 (387.72)
Statistical Analysis 1: Comparison: Dysport® 5U; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 28 days and 112 days
Description: Patients were evaluated for adverse events regarding the use of botulinum toxin, photograph and adverse event questionaire were performed.
Arm/Group | Dysport® 5U/ Botox® 2U
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport® 5U/ Botox® 2U (N=29)
flu (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The field of muscular effects of the studied toxins was objectively measured by EMG and it is not very precise. However, there is no more precise objective measurement to currently evaluate the field effects in muscles than EMG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No